CLINICAL TRIAL: NCT02918812
Title: The Effect of Intracervical Lidocaine Versus Intramuscular Diclofenac for Pain Relief During Hysterosalpingography Among Infertile Women In A Tertiary Hospital In Kano: A Randomized Controlled Trial
Brief Title: Intracervical Lidocaine Versus Intramuscular Diclofenac for Pain Relief in HSG in a Tertiary Hospital in Kano
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayero University Kano, Nigeria (Other)
Responsible Party: Principal Investigator, Sulaiman Muhammaad Daneji, Student, Bayero University Kano, Nigeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ONGDaneji1
Record Dates: First submitted 2016-09-25; First posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Female Infertility of Tubal Origin
Keywords: Hysterosalpingography; Pain relief; Infertility; Intracervical block; Diclofenac
MeSH Terms: conditions — Infertility | interventions — Lidocaine; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intracervical lidocaine (Experimental): This group will comprise of patients that will receive the intracervical block. The study group will receive a total of 60 mg (6 mL) of 1% lidocaine to be injected at four points (12, 4, 6, and 8 o'clock) circumferentially into the cervix (1.5 mL at each point) 5 minutes before proceeding with the hysterosalpingogram.
  Interventions: Drug: Intracervical lidocaine
- Intramuscular Diclofenac (Active Comparator): This group will comprise of patients that will receive intramuscular diclofenac potassium 75mg 30 minutes before proceeding with the hysterosalpingogram.
  Interventions: Drug: Intramuscular Diclofenac

INTERVENTIONS:
Drug: Intracervical lidocaine — Intracervical lidocaine injected at four different points
  Other Names: lignocaine
  Arms: Intracervical lidocaine
Drug: Intramuscular Diclofenac — Intramuscular Diclofenac 30 mins before HSG
  Other Names: Diclofenac sodium; Voltaren
  Arms: Intramuscular Diclofenac

SUMMARY:
This study compares the effect of intracervical block with 1% lidocaine and intramuscular diclofenac 75mg in decreasing pain perception during hysterosalpingography. Half of participants will receive intracervical block with 1% lidocaine, while the other half will receive intramuscular diclofenac 75mg.

DETAILED DESCRIPTION:
Hysterosalpingography (HSG) is a radiographic test to evaluate the contour of the uterine cavity and patency of the fallopian tubes after injection of a radio-opaque dye through the cervix. It is typically performed in the evaluation of infertility or to diagnose uterine anomalies. It is the most common method of tubal evaluation in the developing countries because it is cheap, readily available and requires less expertise. Unfortunately, HSG can cause discomfort or pain for the patient during or after the procedure, and this evokes anxiety and fear for many patients. Up to 72 % of women complain of significant discomfort with this test.

Lidocaine is a local anaesthetic which exerts its effect by altering neuronal depolarization by blocking the sodium channels in the cell membrane, thereby preventing transmission of the sensation of pain to the higher neurons. Lidocaine is commonly used for infiltration and for peripheral nerve blocks if an intermediate duration is required.

Diclofenac is a Non-steroidal anti inflammatory drug that reduce nociception which is related to inflammation and inflammatory mediators whether from trauma

ELIGIBILITY:
Inclusion Criteria:

* All women with infertility who will be undergoing a hysterosalpingography, and must have given consent will be recruited into the study

Exclusion Criteria:

* History of any allergies to local anaesthetics, radio-opaque dye, or anti-inflammatory medications
* All patients with active pelvic inflammatory diseases
* All patients with chronic pelvic pain
* Patients with history of cervical surgery
* Other indications for hysterosalpingography like Ashermans syndrome, congenital uterine anomalies

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analogue Score | Preprocedure and procedure time 0
  A detailed description of the visual analogue scale (VAS) will be given personally to each woman prior to the procedure. The VAS included a 10 cm linear scale on which 0 represents 'no pain' and 10 represents 'worst pain imaginable'. All patients will be asked to grade their perceived lower abdominal pain levels during specified stages of HSG using the VAS as explained to them. The scale will be used at different stages of the procedure: (1) before beginning the procedure; (2) after speculum application but before instrumentation; (3) after the application of the tenaculum and metal cannula and just before the injection of contrast medium; (4) at the end of uterine filling with contrast medium;

SECONDARY OUTCOMES:
patient's satisfaction with pain relief in the two groups using Likert scale | Time Frame: 30 minutes post procedure and 24 hours post procedure
Change in pain score from pre-procedure to 5 and 30 minutes post procedure | 5 minutes and 30 minutes
Change in pain score from pre-procedure to 5 and 24 hours post procedure | 5 minutes and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sulaiman D Muhammad, MBBS, Principal Investigator — Aminu Kano Teaching Hospital
Locations (1):
- Aminu Kano Teaching Hospital, Kano, Kano State, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hamilton M. Infertilty. In Edmonds K (Editor). Dewhurst's Textbook of obstetrics and gynecology. 8th edition. John Wiley and sons ltd 2012 567-79.
- [Background] Hacivelioglu S, Gencer M, Cakir Gungor A, Kosar S, Koc E, Cosar E. Can the addition of a paracervical block to systemic or local analgesics improve the pain perceived by the patient during hysterosalpingography? J Obstet Gynaecol. 2014 Jan;34(1):48-53. doi: 10.3109/01443615.2013.828025. PMID 24359050
- [Background] Chauhan MB, Lakra P, Jyotsna D, Nanda S, Malhotra V. Pain relief during hysterosalpingography: role of intracervical block. Arch Gynecol Obstet. 2013 Jan;287(1):155-9. doi: 10.1007/s00404-012-2515-z. Epub 2012 Aug 28. PMID 22926800
- [Background] Robinson RD, Casablanca Y, Pagano KE, Arthur NA, Bates GW, Propst AM. Intracervical block and pain perception during the performance of a hysterosalpingogram: a randomized controlled trial. Obstet Gynecol. 2007 Jan;109(1):89-93. doi: 10.1097/01.AOG.0000247645.52211.41. PMID 17197592
- [Background] Ahmad G, Duffy J, Watson AJ. Pain relief in hysterosalpingography. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD006106. doi: 10.1002/14651858.CD006106.pub2. PMID 17443612
- [Background] Sinnatamby CS editor. Last's Anatomy: Regional and Applied. 11th Edition. Edinburgh. Churchill Livingstone; 2006. P 311-6.
- [Background] Costello MF, Horrowitz S, Steigrad S, Saif N, Bennett M, Ekangaki A. Transcervical intrauterine topical local anesthetic at hysterosalpingography: a prospective, randomized, double-blind, placebo-controlled trial. Fertil Steril. 2002 Nov;78(5):1116-22. doi: 10.1016/s0015-0282(02)03362-9. PMID 12414003
- [Background] Simpson WL Jr, Beitia LG, Mester J. Hysterosalpingography: a reemerging study. Radiographics. 2006 Mar-Apr;26(2):419-31. doi: 10.1148/rg.262055109. PMID 16549607